CLINICAL TRIAL: NCT04378231
Title: Higher Versus Standard Dose of Amoxicillin-clavulanate in Pediatric Protracted Bacterial Bronchitis: a Randomized Controlled Study.
Brief Title: Higher Versus Standard Dose of Amoxicillin-clavulanate in Pediatric PBB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2018-06-121
Record Dates: First submitted 2020-04-23; First posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Protracted Bacterial Bronchitis
MeSH Terms: interventions — Amoxicillin-Potassium Clavulanate Combination; Amoxicillin; Clavulanic Acid; Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high-dose group (Experimental): patients take dry suspension of amoxicillin clavulanate potassium 45 mg/kg/ time (amoxicillin) orally twice a day, total daily dose not exceeding 2 g, and the course of treatment is two weeks.
  Interventions: Drug: Amoxicillin-Clavulanate 200 Mg-28.5 Mg Oral dry suspension
- standard dose group (Experimental): patients take dry suspension of amoxicillin clavulanate potassium 30 mg/kg/ time (amoxicillin) orally twice a day, total daily dose not exceeding 2 g, and the course of treatment is two weeks.
  Interventions: Drug: Amoxicillin-Clavulanate 200 Mg-28.5 Mg Oral dry suspension

INTERVENTIONS:
Drug: Amoxicillin-Clavulanate 200 Mg-28.5 Mg Oral dry suspension — dry suspension of amoxicillin clavulanate potassium
  Other Names: Amoxicillin and Clavulanate Potassium for Suspension

SUMMARY:
Chronic wet cough is one of the most common symptoms of respiratory diseases in children. Protracted bacterial bronchitis (protracted bacterial bronchitis, PBB) is the most common cause of chronic wet cough in children. Potassium amoxicillin clavulanate is the recommended drug for the treatment of PBB, but there is not enough evidence to date on the dose and course of treatment. investigate the efficacy of different doses of amoxicillin clavulanate sodium in the treatment of chronic bacterial bronchitis in children. The methods of this study are summarized as following:

1. Screening cases of chronic wet cough in children aged 2 to 6 years old who came to our hospital for treatment. Those diagnosed as PBB were included in this study, after obtaining the written informed consent from their parents or guardians.
2. The enrolled patients were randomly divided into high-dose (90mg/kg/d) and standard dose (60mg/kg/d) amoxicillin clavulanate potassium treatment group.
3. Medical history data of enrolled patients and daily cough score data were collected.
4. Assess the cough remission rate within two weeks and recurrence rate within 6 months in both groups.

DETAILED DESCRIPTION:
Chronic cough is one of the common reasons for children seeking medical treatment. In children, chronic cough is associated with impaired quality of life, multiple doctor visits, and adverse effects from inappropriate use of medications. Protracted bacterial bronchitis (PBB) is the most common cause of chronic wet cough in children. Most PBB has a good prognosis, but the persistence of PBB can lead to chronic suppurative lung disease, bronchiectasis and chronic obstructive pneumonia. Therefore, PBB must be timely diagnosed, standardized treatment and strict monitoring to avoid the progression of bronchiectasis and chronic obstructive pulmonary disease.

As in children with chronic wet cough, H. influenzae was the most common pathogen cultured from children with PBB. The other commonly detected bacteria are Strep. pneumoniae and M. catarrhalis and while Staphylococcus aureus. Amoxicillin clavulanate is the most commonly recommended drug for the treatment of PBB, but there is no sufficient evidence for the dose and course of treatment. Therefore, the purpose of this study was to elucidate the optimal dose of amoxicillin clavulanate potassium in the treatment of PBB. It is expected that 100 cases will be included and divided into high-dose group and routine dose group. After grouping, the corresponding dose of amoxicillin clavulanate potassium dry suspension will be prescribed according to the grouping conditions. Patients in high-dose group will receive 90mg/kg/d and the regular dose was 60mg/kg/d, which were taken orally twice a day. Medical history data and daily cough score data of enrolled patients were collected to assess the cough remission rate and recurrence rate within 6 months in both groups.

The research content:

1. Screening cases of chronic wet cough in children aged 2 to 6 years old who came to our hospital for treatment. Those diagnosed with PBB were included in this study after obtaining the written informed consent of their parents or guardians.
2. The enrolled patients were randomly divided into high-dose (90mg/kg/d) and routine dose (60mg/kg/d) amoxicillin clavulanate potassium treatment group.
3. Medical history data of enrolled patients and daily cough score data were collected.
4. Assess the cough remission rate and recurrence rate within 6 months in both groups.

Study design A randomized controlled study for children with protracted bacterial bronchitis

Therapeutic regimens

1. In high-dose group, patients take dry suspension of amoxicillin clavulanate potassium 45 mg/kg/ time (amoxicillin) orally twice a day, total daily dose not exceeding 2 g, and the course of treatment is two weeks.
2. In standard dose group, patients take dry suspension of amoxicillin clavulanate potassium 30 mg/kg/ time (amoxicillin) orally twice a day, total daily dose not exceeding 2 g, and the course of treatment is two weeks.

Effect evaluation

1. Major outcome measure: "cough remission" rate, defined as a more than 75% reduction in verbal category descriptive (VCD) cough score at the end of the study compared to the baseline score at enrollment, or cough cessation for more than 3 days during the study period. The basic score refers to the average VCD of the first two days (-1 and -2 days). The score at the end of the study was the mean score for the first two days (15,16 days) after the 14-day study period.
2. Secondary outcome measures: the absolute change in VCD score and the incidence of adverse events during the study period.

Safety assessment Safety issues will be evaluated before the enrollment and during the follow-up. it mainly included the analysis of meaningful clinical symptoms and adverse events, and the comparison of laboratory tests before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with first-onset PBB
* Subjects and their guardians agree to participate in the study and sign an informed consent

Exclusion Criteria:

* Seriously delayed development of the nervous system;
* With severe underlying diseases: such as severe neuromuscular diseases, immunodeficiency, malnutrition, heart diseases, congenital respiratory system malformation, and other diseases of the heart, brain, liver, kidney and blood system;
* Other diseases that can cause chronic wet cough, including chronic rhinitis, sinusitis, interstitial lung disease, and clinical suspicion of bronchiectasis;
* With poor compliance and expected difficulty in completing the study;
* Other conditions considered inappropriate by the researcher.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
cough remission rate | within two weeks of inclusion
  defined as a more than 75% reduction in VCD cough score at the end of the study compared to the baseline score at enrollment, or cough cessation for more than 3 days during the study period.

SECONDARY OUTCOMES:
the absolute change in VCD score | within two weeks of inclusion
  The basic score refers to the average VCD of the first two days (-1 and -2 days). The score at the end of the study was the mean score for the first two days (15,16 days) after the 14-day study period.
the incidence of adverse events | through their followup completion, an average of half year
  the incidence of any adverse event and severe adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Hai-lin Zhang, MD, Principal Investigator — Second Affiliated Hospital of Wenzhou Medical Universitiy

IPD SHARING:
Plan to Share IPD: No